CLINICAL TRIAL: NCT05148650
Title: Impact of Infusion of Balanced Crystalloid and Colloid Solutions on Haemostasis in Healthy Male Volunteers- a Randomized Controlled Crossover Trial
Brief Title: Impact of Balanced Crystalloid and Colloid Infusion on Haemostasis in Healthy Male Volunteers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Medical University of Silesia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: KNW/0022/KB1/159/II/15161819
Record Dates: First submitted 2021-09-29; First posted 2021-12-08 (Actual); Last update posted 2021-12-08 (Actual); Status verified 2021-09

CONDITIONS: Perioperative Hemorrhage; Dilutional Coagulopathy
Keywords: perioperative hemorrhage; fluid therapy; fluid resuscitation; rotational thromboelastometry; goal-directed therapy; dilutional coagulopathy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Crystalloid infusion (Experimental): Intravenous (IV) transfusions were performed of a 20ml/kg of a balanced crystalloid solution (Optilyte®, Fresenius Kabi). The infusions were performed through an intravenous cannula (18G) inserted into a vein in the antecubital fossa on the non-dominant limb at 1000 ml/h
  Interventions: Diagnostic Test: Standard laboratory coagulation tests and rotational thromboelastometry measurements
- Colloid infusion (Experimental): Intravenous (IV) transfusions were performed of a 20ml/kg of gelatin 26,500 Da (Geloplasma®, Fresenius Kabi). The infusions were performed through an intravenous cannula (18G) inserted into a vein in the antecubital fossa on the non-dominant limb at 1000 ml/h
  Interventions: Diagnostic Test: Standard laboratory coagulation tests and rotational thromboelastometry measurements

INTERVENTIONS:
Diagnostic Test: Standard laboratory coagulation tests and rotational thromboelastometry measurements — Blood for coagulation tests (thromboelastometry, aPTT, PT, INR, fibrinogen concentration, D dimers) and blood morphology was collected just before and immediately after the fluid infusion. With the use of a vacuum system, 20 ml of blood was collected through an IV cannula. The first 5 ml of blood were disposed of due to the possible interference with vascular stasis and fluid infusion on the measurements results.
  Functional tests of coagulation were analysed through ROTEM. ROTEM coagulation analysis was carried out using a ROTEM delta analyzer (Tem Innovations GmbH, Munich, Germany), and assays were allowed to run for 60 minutes. Assays were run immediately after blood sampling to minimize a preanalytical error. Three ROTEM assays were run simultaneously, INTEM, EXTEM, and FIBTEM.

SUMMARY:
The project focuses on perioperative bleeding that requires transfusion of blood products and supplementation of intravascular volume with crystalloids and colloids. The implemented fluid therapy affects coagulation and fibrinolysis, depending on the type of fluid used in an intravenous infusion. Massive haemorrhage significantly impacts the perioperative period and postoperative quality of life and requires individualized therapy, rending the ongoing project relevant from the perspective of the patients.

DETAILED DESCRIPTION:
Perioperative bleeding is a complication that significantly affects postoperative morbidity and quality of life and increases the patient's risk of death. Massive hemorrhage requires individualized therapy, preferably based on international recommendations. It is necessary to transfuse blood and blood products (red blood cells, freshly frozen plasma, platelets, concentrates of coagulation factors) with simultaneous rational supplementation of the intravascular space using crystalloids and colloids. Usually, these are large volumes that are infused over a short time. Proceedings in the operating room and the intensive care unit environment should stabilize the patient's general condition with the lowest possible risk of complications.

However, it has been shown that transfusions are not free from side effects. Transfusions may result not only from "classic" post-transfusion complications (allergic reactions, haemolytic reactions, infections, electrolyte disturbances) but also from iatrogenically generated disorders in the circulatory system (fluid overload), respiratory ( acute lung injury), and hemostasis (risk of hypercoagulability). It is also known that uncontrolled and unbalanced fluid therapy per se may additionally affect the haemodynamic state, haemostasis, and the immune system.

Thromboelastometry (thromboelastography) is becoming the standard of perioperative haemostasis monitoring. It has been documented that it provides more reliable data than standard laboratory tests, such as fibrinogen concentration, activated clotting time (ACT), kaolin-kephalin (aPTT), prothrombin (PT), or INR index. The test can be performed as the so-called point-of-care test (POC), which reduces the waiting time for the result and facilitates goal-directed therapy.

Little is known about the effects of fluid infusion on physiological haemostasis in healthy subjects who do not have a prior bleeding disorder and who are infused with fluids similarly to resuscitation in massive bleeding. Only singular studies in international literature attempted to answer this vital question. Still, the regular progress in the field of fluid therapy makes the obtained data less and less valuable in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers aged 18-30 years
* The American Society of Anaesthesiologists Physical Status (ASA PS) I risk class
* Must be able to give informed consent

Exclusion Criteria:

* Female sex
* Blood type O
* A positive history of any acute diseases in the last four weeks
* Chronic diseases
* Any diagnosed haemostatic disorders
* History of anticoagulation
* Any known bleeding diathesis
* Any pharmacotherapy in the previous week
* Participants were informed about the prohibition of drinking alcohol, excessive exercise, and stress on the day before blood sampling

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2021-02-16 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Rotational thromboelastometry (ROTEM) viscoelastic point-of-care coagulation measurements before and after balanced crystalloid infusion | 60 minutes
  EXTEM, INTEM, FIBTEM assays:
  * A10: clot firmness amplitude measured after 10 minutes (mm)
  * A20: clot firmness amplitude measured after 20minutes (mm)
  * AA: alpha angle (*)
  * CFT: clot forming time (s)
  * CT: clotting time (s)
  * MCE: maximum clot elasticity
  * MCF: maximum clot firmness (mm)
  * ML: maximum lysis (%)
Rotational thromboelastometry (ROTEM) viscoelastic point-of-care coagulation measurements before and after synthetic colloid infusion | 60 minutes
  EXTEM, INTEM, FIBTEM assays:
  * A10: clot firmness amplitude measured after 10 minutes (mm)
  * A20: clot firmness amplitude measured after 20minutes (mm)
  * AA: alpha angle (*)
  * CFT: clot forming time (s)
  * CT: clotting time (s)
  * MCE: maximum clot elasticity
  * MCF: maximum clot firmness (mm)
  * ML: maximum lysis (%)
Standard laboratory tests reporting coagulation status before and after balanced crystalloid infusion | 60 minutes
  * fibrinogen concentration (mg/dl)
  * APTT: activated partial thromboplastin time (s)
  * PT: prothrombin time (s)
  * INR: international normalized ratio
  * PLT: platelet count (10^3/ul)
  * MPV: mean platelet volume (fl)
  * PDW: platelet distribution width (fl)
  * P-LCR: platelet-large cell ratio (%)
Standard laboratory tests reporting coagulation status before and after synthetic colloid infusion | 60 minutes
  * fibrinogen concentration (mg/dl)
  * APTT: activated partial thromboplastin time (s)
  * PT: prothrombin time (s)
  * INR: international normalized ratio
  * PLT: platelet count (10^3/ul)
  * MPV: mean platelet volume (fl)
  * PDW: platelet distribution width (fl)
  * P-LCR: platelet-large cell ratio (%)
Standard laboratory tests reporting fibrinolysis status before and after balanced crystalloid infusion | 60 minutes
  - D-dimer concentration (ug/ml)
Standard laboratory tests reporting fibrinolysis status before and after synthetic colloid infusion | 60 minutes
  - D-dimer concentration (ug/ml)

SECONDARY OUTCOMES:
Safety outcomes after crystalloid and colloid infusion | 28 days
  Assessment of safety and potential of adverse events after fluid infusion

CONTACTS AND LOCATIONS:
Overall Officials: Łukasz J Krzych, Professor, Study Director — Faculty of Medical Sciences in Katowice, Medical University of Silesia; Agnieszka Wiórek, MD, Principal Investigator — Faculty of Medical Sciences in Katowice, Medical University of Silesia
Locations (1):
- Department of Anaesthesiology and Intensive Care, Faculty of Medical Sciences in Katowice, Medical University of Silesia in Katowice, Katowice, Silesian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wiorek A, Mazur PK, Niemiec B, Krzych LJ. Association between Functional Parameters of Coagulation and Conventional Coagulation Tests in the Setting of Fluid Resuscitation with Balanced Crystalloid or Gelatine: A Secondary Analysis of an In Vivo Prospective Randomized Crossover Study. J Clin Med. 2022 Jul 14;11(14):4065. doi: 10.3390/jcm11144065. PMID 35887829